CLINICAL TRIAL: NCT06712589
Title: The Image Characteristics of Adult Appendix on Computed Tomography
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202410072RINB
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Location of Appendix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective analysis of CT images from adult patients who underwent scans for reasons unrelated to appendicitis. The study period will span from January 2010 to August 2024. Through this research, we hope to gain a comprehensive understanding of appendix positioning and compile definitive data on its most common locations.

DETAILED DESCRIPTION:
The investigators conducted a retrospective analysis of CT images from adult patients who underwent scans for reasons unrelated to appendicitis. The study period will span from January 2010 to August 2024. Through this research, we hope to gain a comprehensive understanding of appendix positioning and compile definitive data on its most common locations.

ELIGIBILITY:
Inclusion Criteria:

CT of patients without appendicitis

Exclusion Criteria:

CT of patients with appendicitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigator analyze the location of the normal appendix.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Location of appendix | 1 day
  Analyze the location and categorize to seven groups: preileal, postileal,promontory, pelvic, subcecal, paracecal, retrocecal

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan